CLINICAL TRIAL: NCT00774033
Title: A Randomized Trial Comparing Recell® Autologous Epidermal Cells Harvesting Kits Versus Classic Skin Grafts for the Treatment of Acute Burn in Adults and Children
Brief Title: Epidermal Cells Delivery and Acute Burns
Acronym: ENSEM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients included
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070307
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-03

CONDITIONS: Burn
Keywords: Keratinocytes; Cell spray; Deep partial thickness burns; Full thickness burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment of acute burn in adults and children by epidermal cell spray
  Interventions: Device: autologous epidermal cells harvesting kits
- 2 (Active Comparator): Treatment of acute burn in adults and children by classic skin grafts
  Interventions: Procedure: classic skin grafts

INTERVENTIONS:
Device: autologous epidermal cells harvesting kits — autologous epidermal cells harvesting kits used for the treatment of acute burn
  Other Names: Recell®
  Arms: 1
Procedure: classic skin grafts — classic skin grafts used for the treatment of acute burn
  Arms: 2

SUMMARY:
The aim of the study is to compare results obtained with epidermal cell spray and classic skin grafting for epidermal replacement in acute burns

DETAILED DESCRIPTION:
Comparing the impact in terms of cicatrisation duration and costs between 2 treatments of deep 2nd and 3rd degree burns.

Determine if the costs of the innovating treatment RECELL®, a priori more expensive, are counterbalanced by a shorter cicatrisation duration and an improved evolution versus a conventional strategy.

Give an information about efficiency improvement of RECELL® with additional costs

ELIGIBILITY:
Inclusion Criteria:

* Thermal burns requiring surgical debridement
* Area involved < 1260cm²

Exclusion Criteria:

* local or systemic infection
* conditions that would interfere with wound healing (diabetes, hypertension, inflammatory diseases treated by corticoids)
* hypersensitivity to trypsin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
80% epithelialisation (recipient + owner sites) at one week. Percent epithelialisation at 1, 2 and 6 weeks. | at 1, 2 and 6 weeks

SECONDARY OUTCOMES:
Medical costs at complete epithelialisation | At 6, 12 and 18 months
Post-operative pain | At 6 weeks
Medical assessment of scar quality | at 6 weeks and 6, 12, 18 months
Patient self assessment of scar | At 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GALL, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Trousseau, Paris, France